CLINICAL TRIAL: NCT02038361
Title: Implementation of Innovative Techniques in Routine Diagnosis of Childhood Acute Leukemia: Analysis of Genome and Transcriptome by Micro-array
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-A00263-42; 2013-05 (Other: Assistance Publique Hôpitaux de Marseille)
Record Dates: First submitted 2013-11-25; First posted 2014-01-16 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Acute Leukemia
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- blood sample (Experimental)
  Interventions: Genetic: blood draw

INTERVENTIONS:
Genetic: blood draw

SUMMARY:
Acute leukemias are a heterogeneous group of malignancies characterized by the abnormal proliferation of a cell clone in the bone marrow, having as origin lymphocytic or myeloid lineage. The repertoire of mutations that determine the leukemic transformation, complex and variable depending on the tumor type and progression of the disease, combined in the same cell of balanced and unbalanced chromosomal aberrations, point mutations and epigenetic abnormalities.

The project presented here is part of a comprehensive approach to diagnosis of hematologic malignancies of children. Using comparative genomic hybridization on microarray (or array- CGH) and transcriptome analysis by microarray, two innovative techniques for a comprehensive analysis of the genome and transcriptome , offer new perspectives identifying molecular defects . These techniques provide new elements in the identification of acute leukemia at diagnosis may identify new prognostic factors to optimize the care of patients.

This project involves both the Department of Medical Genetics (Prof. N. LEVY ) regarding the identification of genomic abnormalities associated with childhood leukemia , the Laboratory of Hematology of the Hospital de la Timone ( Prof. Pierre Morange ) in terms of the phenotypic characterization of tumor cells, and the Onco - Hematology Pediatric Department (Prof. Michel Gerard ) which provides diagnosis, treatment , monitoring and the bone marrow of children with hematologic malignancies . The following project is mainly focused on the identification of genomic abnormalities (deletions and duplications) and abnormalities in gene expression to identify a genetic profile ensuring a better classification within the different groups risk .

The project we propose is centered on the identification of genomic abnormalities , changing the number of copies of certain regions of the genome or determining loss of heterozygosity , and the identification of changes in the level of gene expression by using two analytical techniques, comparative genomic hybridization on microarray (or array- CGH) and expression studies with microarrays . The data generated will , for the identification of " molecular signatures " , the classification of patients according to prognosis , variations in treatment response and survival.

The originality of this project lies in the use of these new tools in the diagnosis of hematological malignancies in children. This pilot study will be conducted with commercial Affymetrix , will develop the chips ' processing' , dedicated , enriched probes corresponding to genes involved in leukemogenesis , with high discriminatory power in identifying these signatures.

The data published in the specialized literature from the study of large series of patients show that microarrays provide important information for the diagnosis and therapeutic management of patients. It is for this reason that in the end we hope to integrate these analyzes in routine diagnosis to complement other analyzes ( phenotyping , identification of fusion genes and sequencing) in order to further characterize the abnormal cells leukemia and establish an " identity card of leukemia .

ELIGIBILITY:
Inclusion Criteria:

* patients aged 0-18 years with a diagnosis of acute leukemia

Exclusion Criteria:

* patients without leukemia diagnosis
* patients for which the quantities obtained from DNA and RNA are insufficient

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
identification of genomic abnormalities | 24 months

SECONDARY OUTCOMES:
changing the number of copies of certain regions of the genome or determining loss of heterozygosity | 24 months
identification of changes in the level of gene expression | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille, 80 rue Brochier, 13354 Marseille Cedex 05
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France